CLINICAL TRIAL: NCT04894201
Title: Deep Learning to Summarize Findings in Dental Panoramic Radiographs
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202102018RINB
Record Dates: First submitted 2021-05-09; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Radiography; Digital; Dental Diseases; Dentist-Patient Relations
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients with relevant dental findings
  Interventions: Radiation: Dental Panoramic Radiographs

INTERVENTIONS:
Radiation: Dental Panoramic Radiographs — Exposure to dental panoramic radiographs

SUMMARY:
In this work, the investigators study the application of artificial intelligence systems on dental panoramic images for dental findings. An artificial intelligence system will be learned on an publicly available panoramic image dataset, and test against the investigators' local patient cohort as external test data. The investigators hypothesize the performance would be similar, if not identical to on the public data, and that the investigators' AI system is generalizable.

ELIGIBILITY:
Exclusion Criteria:

* patients under 20 or with primary teeth
* patients with non-removable metal accessory above neck, such as tongue ring, nose ring etc.
* patients with mandible or maxilla deformation

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients with panoramic image exposure and not with exclusion criteria
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve for Receiver Operating Characteristics of Clinical Findings | 1 day
  The investigators use the AI model to infer whether a clinical finding (out of the six type of findings the investigators are interested in) is present in an imaging study from the test set. The result is compared against expert annotation and evaluated for receiver operating characteristics over the whole set. The area under curve will then be calculated and averaged across six type of findings to represent the overall efficacy of the model on detecting findings from panoramic images. From a scale of zero to one, zero is the worst this metric can be and one is the best.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No